CLINICAL TRIAL: NCT01419899
Title: Phase 2/3 Clinical Trial of the Effect of a Brief Intervention on Uptake of Rapid Testing for HIV and Hepatitis C Among Emergency Department Patients
Brief Title: Increasing Viral Testing in the Emergency Department
Acronym: InVITED
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland C. Merchant, MD. MPH, ScD, Associate Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5R21DA28645-2; 5R21DA028645 (NIH)
Record Dates: First submitted 2011-07-06; First posted 2011-08-18 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Drug Use; HIV; Hepatitis C
Keywords: Brief intervention; Rapid testing
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Intervention (Experimental): This arm of the study will receive an assessments survey followed by a brief intervention concerning the relationship between the participants use of drugs and/or sexual risk and rik for HIV and hepatitis C infections. Following the intervention the participants will be offered free rapid testing for HIV and hepatitis C.
  Interventions: Behavioral: Brief motivational intervention
- Standard Care (No Intervention): This arm of the study will receive an assessments survey. Following the assessment the participants will be offered free rapid testing for HIV and hepatitis C.

INTERVENTIONS:
Behavioral: Brief motivational intervention — A 20-30 minute motivational based discussion
  Arms: Brief Intervention

SUMMARY:
The purpose of this study is to determine if a brief intervention delivered to emergency department patients increases the uptake of rapid HIV and hepatitis C testing in comparison to no brief intervention.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient.
* Does not know HIV or hepatitis C status.
* Has an ASSIST V3 score that indicates recent illicit and/or prescription drug use.
* Fluency in English or Spanish.

Exclusion Criteria:

* Critically ill or injured.
* Homicidal and/or suicidal intention.
* Age < 18 years or > 64 years.
* Does not speak English or Spanish.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 398 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The agreement of the participant to be tested for HIV and hepatitis C | Within four hours of being consented into the study
  We will measure the acceptance of free rapid testing for HIV and hepatitis C among the intervention and control groups

SECONDARY OUTCOMES:
Identifying risky sexual behaviors of study participants | Within four hours of being consented into the study
  Identify factors that influence the relationship of BI and risk assessment vs. risk assessment alone on uptake of combined HIV and hepatitis C screening in the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, ScD, Principal Investigator — Brown University; Ted D Nirenberg, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital Emergency Department, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Bernardino VL, Baird JR, Liu T, Merchant RC. Comparison of substance-use prevalence among Rhode Island and The Miriam Hospital Emergency Department patients to state and national general population prevalence estimates. R I Med J (2013). 2014 Apr 1;98(4):30-4. PMID 25830171
- [Derived] Merchant RC, Baird JR, Liu T, Taylor LE, Montague BT, Nirenberg TD. Brief intervention to increase emergency department uptake of combined rapid human immunodeficiency virus and hepatitis C screening among a drug misusing population. Acad Emerg Med. 2014 Jul;21(7):752-67. doi: 10.1111/acem.12419. PMID 25125271
- [Derived] Merchant RC, Baird JR, Liu T, Taylor LE. HCV among The Miriam Hospital and Rhode Island Hospital Adult ED Patients. R I Med J (2013). 2014 Jul 1;97(7):35-9. PMID 24983020